CLINICAL TRIAL: NCT05975879
Title: Multicenter, Prospective, Double-blind, Placebo-controlled, Randomized Study of the Feasibility of Using the Dietary Supplement "ARTNEO®", Capsules for Oral Administration in Patients With Stage II-III Primary Knee Osteoarthritis
Brief Title: A Study of the Feasibility of Using the Dietary Supplement "ARTNEO" in Patients With Osteoathritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NPO Petrovax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Artneo_2021
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2023-07

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis; Knee Osteoarthritis; Knee Arthritis; Knee Discomfort; Knee Pain Swelling; Knee Pain Chronic
Keywords: undenatured type ii collagen; collagen; Boswellia serrata; methylsulfonylmethane; osteoarthritis; knee pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — dimethyl sulfone; Frankincense; Cholecalciferol; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARTNEO (Active Comparator): 1 capsule 1 time per day for 6 months
  Interventions: Dietary Supplement: undenaturated collagen type II, methylsulfonylmethane, boswellia serrata, vitamin D3 (cholecalciferol), vitamin C (ARTNEO)
- Placebo (Placebo Comparator): 1 capsule 1 time per day for 6 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: undenaturated collagen type II, methylsulfonylmethane, boswellia serrata, vitamin D3 (cholecalciferol), vitamin C (ARTNEO) — Release form: capsules with an average weight of 585 mg. Active ingredients: MCM (methylsulfonylmethane) 300 mg, vitamin C (ascorbic acid) 80 mg, boswellia extract (65% boswellic acids) 50.05 mg, undenatured (native) type II collagen 40 mg, vitamin D3 (cholecalciferol) 400 IU.
  Suggested Use: Adults, 1 capsule daily with meals.
  Arms: ARTNEO
Dietary Supplement: Placebo — Release form: capsules with an average weight of 585 mg. No active ingredients.
  Arms: Placebo

SUMMARY:
The goal of this clinical study is to evaluate the effectiveness of the properties that support the functional state of the joints and the safety of the dietary supplement for food ARTNEO®, oral capsules, in patients with stage II-III primary osteoarthritis of the knee joint.

The main questions it aims to answer are:

1. To evaluate the effectiveness of the joint functional state-supporting properties of dietary supplement ARTNEO®, capsules for oral administration, in patients with stage II-III primary osteoarthritis of the knee joint;
2. To evaluate the safety of dietary supplement ARTNEO®, capsules for oral administration, in patients with stage II-III primary osteoarthritis of the knee joint.

Participants will be randomly distributed equally among two groups:

* Group 1 "ARTNEO" (106 people): patients take the study dietary supplement ARTNEO®, 1 capsule 1 time per day for 6 months;
* Group 2 "Placebo" (106 people): patients take placebo 1 capsule 1 time per day for 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed informed consent to participate in the study;
2. Men and women in postmenopause, aged 40-75 years, capable of independent movement, BMI 18-30 kg/m2;
3. Verified primary gonarthrosis according to the American College of Rheumatology criteria at least 6 months before enrollment in the study (in the presence of pain in the knee joint and radiological signs of gonarthrosis in combination with one of the following signs: crepitus in the joint or morning stiffness in the joint for less than 30 min);
4. II-III radiological stage of gonarthrosis according to the Kellgren-Lawrence classification with a predominant lesion of the medial tibiofemoral area of the knee joint;
5. Severity of pain in the assessed knee joint at the time of the screening visit from 40 or more on 100-mm VAS while walking;
6. Ability to understand the rules of the study, willingness to follow them;
7. Willingness to limit the diet (soy, avocado, passion fruit, pineapple, turmeric, linseed, rapeseed, soybean oils, chia seeds, walnuts, decoction of willow bark, pine, wormwood, L-carnitine, etc. should be excluded);
8. Consent of the men during the study and within 30 days after its completion to use the methods of contraception described in the protocol of this study.

Exclusion Criteria:

1. Individual intolerance to the active or excipients of the ARTNEO® dietary supplement (undenatured type II collagen + methylsulfonylmethane + Boswellia serrata extract + vitamin C + Vitamin D3), placebo and the "rescue" drug ibuprofen;
2. Intolerance to eggs, poultry, shellfish;
3. History of trauma or surgery on the target knee joint (other than diagnostic arthroscopy more than 60 days old at study entry), expected surgery (within 6 months following inclusion);
4. Coronary artery bypass grafting in medical history;
5. Diseases, the presence of which, from the point of view of the research physician, puts the patient's health at risk in case of participation in the study or potentially complicates the interpretation of the results of the study (may affect the assessment of endpoints):

   * Known or suspected malignancy at the time of screening or in the previous 2 years, other than completely healed skin cancer in situ;
   * History of gouty arthritis;
   * Malabsorption syndrome, celiac disease, short bowel syndrome, intestinal lymphangiectasia;
   * Peptic ulcer of the stomach and duodenum (in the acute phase or in the acute stage), gastrointestinal bleeding, Crohn's disease, ulcerative colitis at the time of screening or according to medical history for the last 4 months before the screening visit;
   * Hemophilia, hemorrhagic diathesis at the time of screening or according to medical history for the last 4 months before the screening visit, constant use of anticoagulants and antiplatelet agents according to the medical history for the last 4 months before the screening visit;
   * Ischemic heart disease, cerebrovascular disease in the acute stage or decompensation at the time of screening or according to medical history for the last 4 months before the screening visit;
   * Chronic obstructive pulmonary disease (COPD), bronchial asthma according to medical history;
   * Diagnosed moderate or severe chronic renal failure at the time of screening or based on medical history in the last 4 months prior to the screening visit;
   * Moderate to severe hepatic dysfunction as determined by history (any acute liver disease, toxic liver disease, cirrhosis, decompensated liver failure) at the time of screening or from medical history in the last 4 months prior to the screening visit;
   * The presence of rheumatological diseases according to the medical history;
6. Mental and / or neurological diseases with partial or complete loss of legal capacity;
7. Presence or suspicion of drug, alcohol or drug addiction;
8. Intra-articular injection into the target knee joint:

   * Hyaluronates - less than 6 months prior to randomization;
   * Glucocorticosteroids less than 1 month prior to the randomization visit.
   * PRP therapy - less than 6 months prior to randomization
9. The need for constant use of glucocorticoids in any dosage form;
10. Use, including single use, of paracetamol, NSAIDs in any dosage form, and other pain medications within the last 48 hours prior to the randomization visit. Use within 7 days before randomization of certain natural products (such as soy, avocado, passion fruit, pineapple, turmeric, linseed, rapeseed, soybean oils, chia seeds, walnuts, decoction of willow bark, pine, mugwort), L-carnitine;
11. The use of glucosamine or chondroitin during the last 3 months before randomization with a course duration of more than 3 months (if the duration of the course of glucosamine or chondroitin was less than 3 months, then this therapy must be abandoned throughout the study from the moment of the screening visit);
12. Use of ω-3 polyunsaturated fatty acid preparations within 14 days prior to randomization, therapeutic doses of fish oils (≥ 2 g/day) and shark cartilage preparations within 6 months prior to randomization (except vitamin D3);
13. Participation in any clinical trial currently or in the previous 30 days or 5 half-lives (whichever is longer) prior to the Screening visit;
14. History of oral undenatured type II collagen therapy in the last 4 months prior to the screening visit;

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Change in WOMAC-T score | Baseline to month 6
  Change in total Western Ontario and McMaster University Osteoarthritis Index score (WOMAC-T) at Visit 7 (Day 180 ± 4) from start of study dietary supplement/placebo compared to baseline (at Visit 2, Day 1).

SECONDARY OUTCOMES:
Change in the mean score on the subscales of WOMAC | Baseline to months 1, 2, 3, 4, 6
  Change in the mean score on the subscales of Western Ontario and McMaster University Osteoarthritis Index (WOMAC) (pain, stiffness, functional impairment) at Visit 3 (day 30 ± 2), Visit 4 (day 60 ± 2), Visit 5 (day 90 ± 3), Visit 6 (day 120 ± 3) ) and Visit 7 (Day 180 ± 4) compared to baseline (at Visit 2, Day 1);
Change in WOMAC-T score (expt month 6) | Baseline to months 1, 2, 3, 4
  Change in total Western Ontario and McMaster University Osteoarthritis Index score (WOMAC-T) at Visit 3 (day 30 ± 2), Visit 4 (day 60 ± 2), Visit 5 (day 90 ± 3), Visit 6 (day 120 ± 3) compared to basal value (on Visit 2, day 1)
Change in KOOS | Baseline to months 1, 2, 3, 4, 6
  Changes in target joint functional state assessment according to Knee injury and Osteoarthritis Outcome Score (KOOS) at Visit 3 (day 30 ± 2), Visit 4 (day 60 ± 2), Visit 5 (day 90 ± 3), Visit 6 (day 120 ± 3) and Visit 7 (day 180 ± 4) compared to baseline (at Visit 2, day 1);
Ibuprofen intake | Baseline to month 6
  Cumulative oral dose of ibuprofen since day 1 (Visit 2, day 1) and number of patients (%) reporting ibuprofen use;
Drop-out number | Baseline to month 6
  The number of patients dropping out (%) due to the need to prescribe non-steroidal anti-inflammatory drugs (NSAIDs) and other pain medications (with the exception of the drug "rescue" ibuprofen in the doses established by the protocol) or the need to increase the dose allowed under the protocol (more than 1200 mg / day) of ibuprofen;
EQ-5D assessment | Baseline to month 6
  European Quality of Life Questionnaire (EQ-5D) Health Assessment from Baseline (Visit 2, Day 1) at Visit 3 (Day 30 ± 2), Visit 4 (Day 60 ± 2), Visit 5 (Day 90 ± 3), Visit 6 (day 120 ± 3) and Visit 7 (day 180 ± 4)
Pain VAS assessment | Baseline to month 1, 2, 3, 4, 6
  Pain assessment in the target knee on 100 mm visual analog scale (VAS) relative to baseline (Visit 2, Day 1) at Visit 3 (Day 30 ± 2), Visit 4 (Day 60 ± 2), Visit 5 (day 90 ± 3), Visit 6 (day 120 ± 3) and Visit 7 (day 180 ± 4)

OTHER OUTCOMES:
Synovitis severity | Baseline to month 6
  Assessing the severity of synovitis according to the results of ultrasound examination of the target knee joint from the basal level (Visit 2, Day 1) at Visit 7 (Day 180 ± 4)
14-day pain VAS assessment | Baseline to day 14
  Assessment of the severity of pain when walking in the target knee joint on a 100-mm visual analog scale (VAS) relative to the basal level (Visit 2, day 1) on day 14±1.

CONTACTS AND LOCATIONS:
Overall Officials: Ludmila Alekseeva, MD, Principal Investigator — FSBSI "Research Institute of Rheumatology named after V.A. Nasonova"
Locations (11):
- Russia (11):
  - NIMK Vashe Zdorovie LLC, Kazan'
  - Federal State Budgetary Scientific Institution "Research Institute of Rheumatology named after V.A. Nasonova", Moscow
  - Pirogov Russian National Research Medical University, Moscow
  - Research Center Eco-Safety LLC, Saint Petersburg
  - Energiia Zdoroviya LLC, Saint Petersburg
  - "Medical Sanitary Unit No. 157" LLC, Saint Petersburg
  - Zvezdnaya Clinic LLC, Saint Petersburg
  - Meili LLC, Saint Petersburg
  - State Health Institution "Tula Regional Clinical Dermatovenerologic Dispensary", Tula
  - Ulyanovsk Regional Clinical Hospital, Ulyanovsk
  - Private educational institution of additional professional education 'Institute for advanced training and professional retraining of personnel, Yaroslavl

IPD SHARING:
Plan to Share IPD: No